CLINICAL TRIAL: NCT01006083
Title: Impact of Continued Use of Clopidogrel and / or Aspirin on Outcomes in Patients Undergoing Lumbar Spine Surgery. A Prospective Observational Study
Brief Title: Antiplatelet Therapy Continuation in Spine Surgery - Its Effect on Postoperative Morbidity and Mortality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof. Idit Matot, Department of Anesthesiology & Intensive Care, Tel Aviv Sourasky medical center
Other Study IDs: TASMC-09-IM-0540-CTIL
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Hemorrhage; Cerebrovascular Accident; Myocardial Infarction; Pulmonary Embolism; Deep Vein Thrombosis
Keywords: Aspirin; Plavix; antiplatelet therapy; Hemorrhage; ischemic events
MeSH Terms: conditions — Hemorrhage; Stroke; Myocardial Infarction; Pulmonary Embolism; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Low-risk patients, not on APAs: Patients not at risk of coronary and/or cerebrovascular disease, and not consuming APAs
- High-risk patients, not on APAs: Patients at high risk for cardio/cerebrovascular disease (diabetes mellitus, cigarette smoking, hypercholesterolemia, hypertension, morbid obesity), but not taking APAs.
- APA for primary prevention: High-risk patients with cardiovascular risk factors (as above), in whom APA is prescribed as primary prevention of coronary artery disease (CAD).
- APA for secondary prevention: Patients with a history of a coronary syndrome (stable/unstable angina); MI; transient ischemic attack (TIA)/stroke; severe carotid artery stenosis/stenting; or peripheral vascular disease, on APAs for secondary prevention.

SUMMARY:
The objective of this study is to evaluate the safety of antiplatelet (APA)therapy continuation in patients undergoing lumbar spine surgery (laminectomy, discectomy and foraminotomy), and to gather evidence-based data regarding postoperative outcomes potentially related to APA management.

DETAILED DESCRIPTION:
BACKGROUND Antiplatelet agents (APAs) are widely prescribed for coronary stenting, primary and secondary prevention of cerebrovascular and coronary artery disease. Dual antiplatelet therapy (aspirin/plavix) has become the mainstay antiplatelet treatment strategy for the prevention of stent thrombosis. Maintaining antiplatelet therapy until the end of the indicated period is crucial for the success of coronary stents. Premature discontinuation of antiplatelet therapy markedly increases the risk of stent thrombosis, a catastrophic event that frequently leads to myocardial infarction (MI), with a death rate of 20-40%. Aspirin is commonly prescribed for lifetime in patients at increased atherothrombotic risk, whereas Plavix is regarded as mandatory until the coronary stents are fully endothelialized, which takes 4-6 weeks for bare metal stents and up to 1 yr for drug-eluting stents. And yet, within the first year after stenting, approximately 5% of patients who have undergone percutaneous coronary interventions (PCIs) will require noncardiac surgery, thus raising dilemmas of APA management: stopping APA treatment before operation to avoid bleeding while risking postoperative stent thrombosis versus maintaining APA therapy perioperatively thus risking extensive blood loss but limiting the risks of postoperative ischemic events.

Current recommendations are that aspirin should not be discontinued pre-operatively, with the exception of brain surgery and certain urological operations in which bleeding may be difficult to control and is therefore life threatening.

The continued use of plavix during the perioperative period significantly increases intraoperative blood loss, re-operations for the control of hemorrhage and transfusions, but does not affect morbidity, mortality, or surgical outcomes.

Most guidelines recommend to postpone invasive procedures until the end of the indication for plavix. Only vital or emergency surgery should be performed on full antiplatelet therapy, with the exception of procedures in which even a small hemorrhage may have disastrous consequences (e.g. intracranial surgery, spinal surgery in the medullary canal, surgery of the posterior chamber of the eye), or procedures involving massive bleeding.

Evidence-based data are needed to guide management of patients in whom early antiplatelet withdrawal is being considered (e.g. those who require non-cardiac surgery). Several studies have been conducted in orthopedic and cardiac surgery, however, to the best of our knowledge, not in spine surgery. This type of surgery might often be semi-urgent and postponing surgery for long time may be problematic.

This prospective, observational study is designed to evaluate the safety of APA therapy continuation in patients admitted for lumbar spine surgery.

METHODS

Study design The study will be conducted as an observational one. An informed consent will be obtained from all patients matching the above criteria. Diuretics and oral hypoglycemics will be discontinued the day prior to surgery, as dictated by the routines in our patients. Antiplatelet therapy will be continued as commonly practiced in these procedures. Any deviation from this protocol will be documented. Throughout the postoperative period study patients will be observed for any bleeding- or thrombosis-related events, and relevant perioperative data will documented (see "patient monitoring & assessment").

Peri-operative management Anesthetic and surgical management, including management of surgical hemorrhage or any other hemodynamic event will adhere to standard practice. Postoperatively, study patients will be transferred to the post-anesthesia care unit and later to the neurosurgery department, unless otherwise indicated. In the postoperative period, departmental routines will guide blood product transfusions, pain management, fluid regimens and medications administered.

Patient monitoring & assessment

Patients will be allocated into 4 groups:

1. Patients not at risk of coronary and/or cerebrovascular disease, and not taking APAs.
2. Patients at high risk for cardio/cerebrovascular disease (diabetes mellitus, cigarette smoking, hypercholesterolemia, hypertension, morbid obesity), but not taking APAs.
3. High-risk patients with cardiovascular risk factors (as above), in whom APA is prescribed as primary prevention of coronary artery disease (CAD).
4. Patients with a history of a coronary syndrome (stable/unstable angina); MI; transient ischemic attack (TIA)/stroke; severe carotid artery stenosis/stenting; or peripheral vascular disease, on APAs for secondary prevention.

For each consented patient included in the study we will record demographics and medical history ; chronic medications ; detailed cardiovascular history ; neurological examination ; APA-related data: type and dose of APA taken; indication ; Intra-operative data ; and perioperative complications.

Outcome measures

1. Primary outcomes: hemorrhagic, thrombotic, and neurological complications Include any complication, morbidity or death potentially caused by continuation (e.g., direct or indirect hemorrhage; hemorrhagic CVA) or withdrawal of APA therapy (e.g., MI; PE; ischemic CVA; DVT; etc.), occurring until discharge, or within 30 postoperative days. Neurological complications may be related to surgery; bleeding; thrombosis; other, and will be classified accordingly.
2. Secondary outcomes Include: re-intubations; transfer to ICU; length of stay (LOS); re-admissions within 7 / 30 days; major morbidity or death 30 and 60 days postoperatively.

Study size The study is expected to last 2 years, and to include approximately 200 patients.

REFERENCES

1. Anderson, J.L., et al., ACC/AHA 2007 guidelines for the management of patients with unstable angina/non-ST-Elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non-ST-Elevation Myocardial Infarction) developed in collaboration with the American College of Emergency Physicians, the Society for Cardiovascular Angiography and Interventions, and the Society of Thoracic Surgeons endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic Emergency Medicine. J Am Coll Cardiol, 2007. 50(7): p. e1-e157.
2. Fox, K.A., et al., Benefits and risks of the combination of clopidogrel and aspirin in patients undergoing surgical revascularization for non-ST-elevation acute coronary syndrome: the Clopidogrel in Unstable angina to prevent Recurrent ischemic Events (CURE) Trial. Circulation, 2004. 110(10): p. 1202-8.
3. Hirsch, A.T., et al., ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation, 2006. 113(11): p. e463-654.
4. Keller, T.T., A. Squizzato, and S. Middeldorp, Clopidogrel plus aspirin versus aspirin alone for preventing cardiovascular disease. Cochrane Database Syst Rev, 2007(3): p. CD005158.
5. Smith, S.C., Jr., et al., AHA/ACC guidelines for secondary prevention for patients with coronary and other atherosclerotic vascular disease: 2006 update: endorsed by the National Heart, Lung, and Blood Institute. Circulation, 2006. 113(19): p. 2363-72.
6. Weitz, J.I., J. Hirsh, and M.M. Samama, New antithrombotic drugs: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest, 2008. 133(6 Suppl): p. 234S-256S.
7. Grines, C.L., et al., Prevention of premature discontinuation of dual antiplatelet therapy in patients with coronary artery stents: a science advisory from the American Heart Association, American College of Cardiology, Society for Cardiovascular Angiography and Interventions, American College of Surgeons, and American Dental Association, with representation from the American College of Physicians. Circulation, 2007. 115(6): p. 813-8.
8. Iakovou, I., et al., Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA, 2005. 293(17): p. 2126-30.
9. Patrono, C., et al., Antiplatelet drugs: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest, 2008. 133(6 Suppl): p. 199S-233S.
10. Pfisterer, M., et al., Late clinical events after clopidogrel discontinuation may limit the benefit of drug-eluting stents: an observational study of drug-eluting versus bare-metal stents. J Am Coll Cardiol, 2006. 48(12): p. 2584-91.
11. Ong, A.T., et al., Late angiographic stent thrombosis (LAST) events with drug-eluting stents. J Am Coll Cardiol, 2005. 45(12): p. 2088-92.
12. Schouten, O., J.J. Bax, and D. Poldermans, Management of patients with cardiac stents undergoing noncardiac surgery. Curr Opin Anaesthesiol, 2007. 20(3): p. 274-8.
13. Laffey, J.G., J.F. Boylan, and D.C. Cheng, The systemic inflammatory response to cardiac surgery: implications for the anesthesiologist. Anesthesiology, 2002. 97(1): p. 215-52.
14. Priebe, H.J., Triggers of perioperative myocardial ischaemia and infarction. Br J Anaesth, 2004. 93(1): p. 9-20.
15. Ho, P.M., et al., Incidence of death and acute myocardial infarction associated with stopping clopidogrel after acute coronary syndrome. JAMA, 2008. 299(5): p. 532-9.
16. Ferrari, E., et al., Coronary syndromes following aspirin withdrawal: a special risk for late stent thrombosis. J Am Coll Cardiol, 2005. 45(3): p. 456-9.
17. Sharma, A.K., et al., Major noncardiac surgery following coronary stenting: when is it safe to operate? Catheter Cardiovasc Interv, 2004. 63(2): p. 141-5.
18. Chassot, P.G., A. Delabays, and D.R. Spahn, Perioperative antiplatelet therapy: the case for continuing therapy in patients at risk of myocardial infarction. Br J Anaesth, 2007. 99(3): p. 316-28.
19. Chu, M.W., et al., Does clopidogrel increase blood loss following coronary artery bypass surgery? Ann Thorac Surg, 2004. 78(5): p. 1536-41.
20. Douketis, J.D., et al., The perioperative management of antithrombotic therapy: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest, 2008. 133(6 Suppl): p. 299S-339S.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years old,
* Undergoing elective or urgent spinal surgery,
* Included are procedures aimed to decompress the spinal canal in the lumbar region due to a degenerative disease, i.e., laminectomy, discectomy and foraminotomies.

Exclusion Criteria:

* Patients with an infectious disease, tumor resection, trauma cases, or
* Patients requiring lumbar fixation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for lumbar laminectomy, discectomy or foraminotomy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative hemorrhagic, thrombotic, and neurological complications | 60 days

SECONDARY OUTCOMES:
length of stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel